CLINICAL TRIAL: NCT04629118
Title: Intervention With Selution SLR™ Agent Balloon for Endovascular Latent Limus Therapy for Failing AV Fistulas (ISABELLA) Trial
Acronym: ISABELLA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/2782
Record Dates: First submitted 2020-11-08; First posted 2020-11-16 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Arteriovenous Fistula; Dialysis Access Malfunction
Keywords: Drug-Coated Balloons; Sirolimus; Arteriovenous Fistula; Fistuloplasty
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Selution SLR™ 018 Drug Eluting Balloon: Subjects will undergo fistuloplasty with the study device - Selution SLR™ 018 Drug Eluting Balloon
  Interventions: Device: Selution SLR™ 018 Drug Eluting Balloon

INTERVENTIONS:
Device: Selution SLR™ 018 Drug Eluting Balloon — Target lesion will be pre-dilated with high pressure non-compliant balloon, then treated with SELUTION SLR™ 018 DEB Balloon.
  Other Names: Sirolimus DEB

SUMMARY:
The most common problem with haemodialysis arteriovenous fistulas (AVF) and arterio-venous grafts (AVG) is stenosis, which can lead to inadequate dialysis, and eventual access thrombosis. Conventional plain old balloon angioplasty (CBA) is associated with high recurrence rates of stenosis and repeated interventions. The advent of successful drug-eluting technology in the treatment of the coronary vascular bed and subsequent positive accumulating evidence in the peripheral arterial circulation has prompted the use of drug coated balloons (DCB) in the access fistula circuit for venous stenosis and in-stent restenosis. Recent studies suggest that DCBs may significantly reduce re-intervention rates on native and recurrent lesions. The restenosis process is in part or in whole the result of neo-intimal hyperplasia (NIH) and NIH is considered the main culprit in access circuit target lesion stenosis. NIH is the blood vessel's healing response to the barotrauma from the angioplasty process. A critical component of NIH is the cellular proliferative stage with mononuclear leucocytes identified as the primary inflammatory cell type involved. The rationale for drug elution is to block the NIH response with an anti-metabolite such as paclitaxel. It is important to emphasize that the role of drug elution in the treatment of vascular stenosis is not to obtain a good haemodynamic and luminal result but to preserve a good result obtained during POBA from later restenosis due to NIH and minimise reinterventions and readmissions to hospital for what is a frail population of patients.

A meta-analysis performed by Khawaja et al. seemed to suggest that DCBs conferred some benefit in terms of improving target lesion primary patency (TLPP) in AVFs. An updated meta-analysis performed by our own institution recently reinforced that DCB appears to be a better and safe alternative to CBA in treating patients with stenosis within all haemodialysis circuits (fistulas and grafts) based on 6- and 12-months primary patency and increased intervention free period 5. However, this was not reflected in the largest RCT to date of DCB vs CBA in AVF with no superior target lesion patency demonstrated at six months and one and two years follow-up. Another recent meta-analysis found paclitaxel-coated balloons (PCB) showed no statistically significant improvement over conventional balloons in decreasing fistula stenosis in randomized controlled trials but were significant for cohort studies. Hence this shows the heterogeneity of the available data in the literature and the result is dependent on what studies you include in the review. Another reason why the outcome data is variable is that the high-speed blood flow in dialysis access circuits washes a large amount of the paclitaxel away from the target lesion soon after application. A measurement in swine showed that only 20%-30% of paclitaxel was taken up into the coronary artery wall in vivo 15-25minutes after PCB application.

Furthermore, recent attention has been drawn to a possible increase in late mortality signal and lower amputation free survival in patients receiving DCB treatment with paclitaxel for peripheral arterial disease, although this suggestion has not been demonstrated in the data of DCB within the fistula circuit either at 1 or 2 years. In light of these concerns, attention has turned away recently from paclitaxel-based technologies to sirolimus coated platforms. Sirolimus, like paclitaxel, is a potent antiproliferative agent, which has been found to prevent restenosis in the coronary bed and more recently in the peripheral vasculature but to date has not been studied in AVF circuits The aims of the study is to determine the safety and efficacy of the MedAlliance SELUTION SLR 018™ DEB in the treatment of failing AV fistula due to conduit stenosis in patients undergoing renal dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥21 years and ≤90 years
* Native AVF was created more than 2 months prior to the index procedure and had undergone 10 or more haemodialysis sessions utilising two needles
* Target lesion location has to be located between the anastomoses to the auxiliary-subclavian vein junction, as defined by insertion of the cephalopods vein
* On initial fistulogram, target lesion stenosis has to be >50% on angiographic assessment and in keeping with the clinical indicator for intervention
* Stenosis had to be < 12cm in length (to allow for potential treatment with one DEB (length 15cm) only)
* Stenosis had to be initially treated successfully with a high-pressure plain balloon prior to DEB treatment as defined by:- (A) No clinically significant dissection (flow limiting) (B) No extravasated requiring treatment/Stenting (C) Residual stenosis ≤30% by angiographic measurement (D) Ability to completely efface the lesion waist using the pre-dilation CBA
* No more than one additional ("non-target") lesion in the access circuit that had to be also successfully treated (≤30% residual stenosis) before drug elation. Separate lesion was defined by at least 3cm in distance from the target lesion
* Reference vessel diameters allowed are 4mm - 7mm

Exclusion Criteria:

* Women who are pregnant, lactating or planning on becoming pregnant during study
* Subject has more than two lesions in the access circuit
* Subject had a secondary non-target lesion that could not be successfully treated
* Sepsis or active infection
* Asymptomatic target lesions
* A thrombosis access or an access with thrombosis treated ≤30 days prior to the index procedure
* Pseudoaneurysm in proposed target lesion area
* Surgical revision of the access site performed, planned or expected ≤3 months before or after the index procedure
* Patients who is taking immunosuppressive therapy or are routinely taking ≥15mg of prednisone per day
* Currently participating in another investigational drug, biologic, or device study involving Sirolimus or Paclitaxel
* Contraindication to aspirin or clopidogrel usage
* Mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study, or language barrier such that the subject is unable to give informed consent.
* Uncooperative attitude or potential for non-compliance with the requirements of the protocol making study participation impractical
* Where final angioplasty treatment requires a stent or drug eluting balloon >8mm in diameter
* Metastatic cancer or terminal medical condition
* Blood coagulation disorders
* Limited life expectancy (<12 months)
* Allergy or other known contraindication to iodinated media contrast, heparin, or Sirolimus

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 patients with failing dialysis access treated with SELUTION SLR and meet inclusion/exclusion criteria will be enrolled for study
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-10-27 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Primary Patency | 6 months post-index procedure
  Defined as patency with no re-intervention to the area treated by SELUTION SLR™ DEB and a duplex-defined stenosis within the index-treated segment of <50%. TLPP ends when any of the following occur:- 1) clinically driven re-intervention to the treated segment, 2) thrombotic occlusions that includes the treatment segment, 3) surgical intervention that excludes the treatment segment from the access circuit, 4) abandonment of the AVF due to an inability to treat the target lesion, 5) duplex finding of more than 50% stenosis.
Freedom from adverse events | 30 days post-index procedure
  Freedom from events including thrombosis, life-threatening events or those resulting in death, requiring hospitalisation, resulting in permanent disability, requiring intervention to prevent permanent impairment.

SECONDARY OUTCOMES:
Freedom from any serious adverse event(s) involving the AV access circuit or the patient | 3 and 6 months post-index procedure
Target Lesion Primary Patency and Access circuit primary patency | 3 months post index procedure
  Defined as patency with no re-intervention to the area treated by SELUTION SLR™ DEB and a duplex-defined stenosis within the index-treated segment of <50%. TLPP ends when any of the following occur:- 1) clinically driven re-intervention to the treated segment, 2) thrombotic occlusions that includes the treatment segment, 3) surgical intervention that excludes the treatment segment from the access circuit, 4) abandonment of the AVF due to an inability to treat the target lesion, 5) duplex finding of more than 50% stenosis.
Device Success | Intra-operative
  Successful balloon inflation of the SELUTION catheter for more than 2 minutes and retrieval of the catheter
Anatomical Success | Immediately post-op
  <30% residual stenosis diameter measured immediately after an angioplasty
Clinical Success | 1 week post-index procedure
  Improvement from baseline in the clinical or hemodynamic parameter (e.g. blood flow, venous pressure) that was the initial indicator of fistula dysfunction and the resumption of normal hemodialysis for a minimum of at least 1 session following the procedure
Need for open revision surgery | 2 years post-index procedure
Secondary patency | 3 months and 6 months post-index procedure
  Interval after intervention until access circuit is abandoned, including reinterventions to reestablish access flow.
Access circuit thrombosis | 2 years post-index procedure
Number of interventions required to maintain access circuit patency | 3 and 6 months post-index procedure
Mortality rate | 3 and 6 months post-index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Tjun Yip Tang, Principal Investigator — Singapore General Hospital; Tze Tec Chong, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Troisi N, Frosini P, Somma C, Romano E, Guidotti A, Dattolo PC, Ferro G, Chisci E, Michelagnoli S. Drug-coated balloons reduce the risk of recurrent restenosis in arteriovenous fistulas and prosthetic grafts for hemodialysis. Int Angiol. 2018 Feb;37(1):59-63. doi: 10.23736/S0392-9590.17.03886-X. Epub 2017 Nov 10. PMID 29125264
- [Background] Kennedy SA, Mafeld S, Baerlocher MO, Jaberi A, Rajan DK. Drug-Coated Balloon Angioplasty in Hemodialysis Circuits: A Systematic Review and Meta-Analysis. J Vasc Interv Radiol. 2019 Apr;30(4):483-494.e1. doi: 10.1016/j.jvir.2019.01.012. Epub 2019 Mar 8. PMID 30857987
- [Background] Roy-Chaudhury P, Sukhatme VP, Cheung AK. Hemodialysis vascular access dysfunction: a cellular and molecular viewpoint. J Am Soc Nephrol. 2006 Apr;17(4):1112-27. doi: 10.1681/ASN.2005050615. PMID 16565259
- [Background] Khawaja AZ, Cassidy DB, Al Shakarchi J, McGrogan DG, Inston NG, Jones RG. Systematic review of drug eluting balloon angioplasty for arteriovenous haemodialysis access stenosis. J Vasc Access. 2016 Mar-Apr;17(2):103-10. doi: 10.5301/jva.5000508. Epub 2016 Feb 5. PMID 26847736
- [Background] Trerotola SO, Saad TF, Roy-Chaudhury P; Lutonix AV Clinical Trial Investigators. The Lutonix AV Randomized Trial of Paclitaxel-Coated Balloons in Arteriovenous Fistula Stenosis: 2-Year Results and Subgroup Analysis. J Vasc Interv Radiol. 2020 Jan;31(1):1-14.e5. doi: 10.1016/j.jvir.2019.08.035. Epub 2019 Nov 6. PMID 31706886
- [Background] Abdul Salim S, Tran H, Thongprayoon C, Fulop T, Cheungpasitporn W. Comparison of drug-coated balloon angioplasty versus conventional angioplasty for arteriovenous fistula stenosis: Systematic review and meta-analysis. J Vasc Access. 2020 May;21(3):357-365. doi: 10.1177/1129729819878612. Epub 2019 Oct 9. PMID 31595799
- [Background] Kelsch B, Scheller B, Biedermann M, Clever YP, Schaffner S, Mahnkopf D, Speck U, Cremers B. Dose response to Paclitaxel-coated balloon catheters in the porcine coronary overstretch and stent implantation model. Invest Radiol. 2011 Apr;46(4):255-63. doi: 10.1097/RLI.0b013e31820577df. PMID 21285890
- [Background] Katsanos K, Spiliopoulos S, Kitrou P, Krokidis M, Karnabatidis D. Risk of Death Following Application of Paclitaxel-Coated Balloons and Stents in the Femoropopliteal Artery of the Leg: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Am Heart Assoc. 2018 Dec 18;7(24):e011245. doi: 10.1161/JAHA.118.011245. PMID 30561254
- [Background] Katsanos K, Spiliopoulos S, Kitrou P, Krokidis M, Paraskevopoulos I, Karnabatidis D. Risk of Death and Amputation with Use of Paclitaxel-Coated Balloons in the Infrapopliteal Arteries for Treatment of Critical Limb Ischemia: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Vasc Interv Radiol. 2020 Feb;31(2):202-212. doi: 10.1016/j.jvir.2019.11.015. Epub 2020 Jan 15. PMID 31954604
- [Background] Cao Z, Li J, Zhang T, Zhao K, Zhao J, Yang Y, Jiang C, Zhu R, Li Z, Wu W. Comparative Effectiveness of Drug-Coated Balloon vs Balloon Angioplasty for the Treatment of Arteriovenous Fistula Stenosis: A Meta-analysis. J Endovasc Ther. 2020 Apr;27(2):266-275. doi: 10.1177/1526602820902757. Epub 2020 Feb 11. PMID 32043432
- [Background] Tang TY, Choke EC, Walsh SR, Tiwari A, Chong TT. What Now for the Endovascular Community After the Paclitaxel Mortality Meta-Analysis: Can Sirolimus Replace Paclitaxel in the Peripheral Vasculature? J Endovasc Ther. 2020 Feb;27(1):153-156. doi: 10.1177/1526602819881156. Epub 2019 Oct 14. No abstract available. PMID 31608741
- [Background] Ali RM, Abdul Kader MASK, Wan Ahmad WA, Ong TK, Liew HB, Omar AF, Mahmood Zuhdi AS, Nuruddin AA, Schnorr B, Scheller B. Treatment of Coronary Drug-Eluting Stent Restenosis by a Sirolimus- or Paclitaxel-Coated Balloon. JACC Cardiovasc Interv. 2019 Mar 25;12(6):558-566. doi: 10.1016/j.jcin.2018.11.040. PMID 30898253
- [Background] Tang TY. How Low Can You Go? SELUTION SLR™ Tibial Artery Drug-Coated Balloon Angioplasty in the Setting of CLTI Conference Proceedings 2020; Leipzig Interventional Course (LINC), Leipzig, Germany